CLINICAL TRIAL: NCT00134628
Title: Hyperbaric Oxygen Radiation Tissue Injury Study - Project HORTIS
Brief Title: Study to Determine if Hyperbaric Oxygen Therapy is Helpful for Treating Radiation Tissue Injuries
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinued cystitis study due to poor recruitment. To continue the trial under these circumstances is considered non-viable.
Sponsor: National Baromedical Services (Other)
Responsible Party: Principal Investigator, Dick Clarke, President, National Baromedical Research Foundation, National Baromedical Services
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Project HORTIS; ISRCTN85456814
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2012-02

CONDITIONS: Radiation Injuries
Keywords: Hyperbaric Oxygenation; Radiation injuries; Prophylaxis; Proctitis; Cystitis; Enteritis; Osteoradionecrosis
MeSH Terms: conditions — Radiation Injuries; Proctitis; Cystitis; Enteritis; Osteoradionecrosis | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Hyperbaric Oxygen Therapy
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- B (Sham Comparator): Normal Air
  Interventions: Procedure: Sham treatment

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — HBO at 2.0 ATA
  Arms: A
Procedure: Sham treatment — Normal air under pressure (1.1 ATA)
  Arms: B

SUMMARY:
The principle objective of this research is to more precisely determine the degree of benefit that hyperbaric oxygen therapy affords in the treatment of late radiation tissue injury.

The study has eight* components. Seven involve the evaluation of established radionecrosis at varying anatomic sites (mandible, larynx, skin, bladder, rectum, colon, and gyn). The eighth will investigate the potential of hyperbaric oxygen (HBO) therapy to prophylax against late radiation tissue injury.

*(One of the arms, HORTIS IV - Proctitis has been closed to further patient recruitment. This decision was based on an interim statistical analysis which generated sufficient evidence to support closing down this arm of HORTIS.)

DETAILED DESCRIPTION:
Radiation therapy is a key component of the control and eradication of malignant disease. Adequate tumoricidal doses may, however, result in damage to surrounding healthy tissue. Therapeutic radiation injuries to non-target tissues can be divided into acute, sub-acute, and delayed complications. Acute injuries are considered a direct cellular toxicity, self-limiting, and in most cases successfully managed symptomatically. Sub-acute injuries are typically identifiable in only a few organ systems, e.g., radiation pneumonitis. These, too, are generally limited but occasionally evolve to late complications. Late changes occur several months to many years after completing radiotherapy.

The etiology of radiation's late effects to normal tissue (LENT) varies somewhat between organ systems. Its hallmark, however, is one of culminating in an obliterative endarteritis, and local hypoxia.

The incidence of LENT is related to both total radiation exposure and the length of time a patient is out from completing radiotherapy. The higher the dose, the longer the interval from exposure, the greater the risk. In many cases, resulting radionecrotic lesions seriously impair form and function, and require extensive surgical correction or repair. Such surgery is fraught with complications, hence the inclusion of a "prophylactic" hyperbaric oxygen arm. A disturbing degree of mortality further complicates the development of LENT.

Hyperbaric oxygen has been utilized in the treatment of radiation tissue injury for several decades. Most of the supportive basic science and clinical evidence stems from the management of mandibular osteoradionecrosis. More recently, the use of hyperbaric oxygen has been extended to other anatomic sites. This expanded use is based, in large part, on a presumed common underlying pathophysiology of LENT, regardless of its anatomic location. Supportive clinical evidence for these other sites is limited, however, and in need of a greater degree of scientific scrutiny.

ELIGIBILITY:
Inclusion Criteria:

* Endarteritis
* Hypovascularity
* Diarrhea
* Cramping
* Obstruction
* Stricture
* Pain
* Hemorrhage
* Wall Changes
* Ulceration
* Hypocellularity
* Mucosal thickening
* Vomiting
* Tenesmus
* Constipation
* Perforation
* Fistula
* Obstipation
* Tissue hypoxia

Exclusion Criteria:

* Pregnancy
* Reactive airway disease
* Radiographic evidence of pulmonary blebs or bullae
* Untreated pneumothorax
* Previously documented ejection fraction less than 35%
* History of seizures except childhood febrile seizures
* Cardiovascular instability
* Mechanical ventilator support with the exception of those patients who are immediately (1-5 days) post-operative
* Unable to follow simple commands
* Not orientated to person, place, time
* Participating as a subject in any other medical or biomedical research project; if previously involved as a subject, sufficient time must have elapsed to permit "wash out" of any investigational agent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2001-01; Primary Completion 2011-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
SOMA (Subjective, Objective, Management, Analytic) scale used to determine late effects to normal tissue (LENT) score | pre-treatment, post-treatment (HBO and placebo) and at follow ups at 3 months, 6 months, and 1 year through 5 years

SECONDARY OUTCOMES:
Clinical assessment using one of the following criteria: | post-treatment (HBO and placebo) and at follow ups at 3 months, 6 months, and 1 year through 5 years
Healed | post-treatment (HBO and placebo) and at follow ups at 3 months, 6 months, and 1 year through 5 years
Modestly improved (< 50% lesion resolution) | post-treatment (HBO and placebo) and at follow ups at 3 months, 6 months, and 1 year through 5 years
Not improved | post-treatment (HBO and placebo) and at follow ups at 3 months, 6 months, and 1 year through 5 years
Other (e.g. lesion recurrence, lesion size progression) | post-treatment (HBO and placebo) and at follow ups at 3 months, 6 months, and 1 year through 5 years
Significant Improvement (>50% lesion resolution) | post-treatment (HBO and placebo) and at follow ups at 3 months, 6 months, and 1 year through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dick Clarke, CHT, Principal Investigator — National Baromedical Services
Locations (7):
- Palmetto Health Richland, Columbia, South Carolina, United States
- Australia (2):
  - Wesley Medical Center, Brisbane, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
- Instituto Nacional de Cancerologica, Mexico City, Mexico
- South Africa (2):
  - University of Stellenbosch, Cape Town
  - University of Pretoria Medical Center, Pretoria
- Istanbul University Medical Center, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Curi MM, Dib LL. Osteoradionecrosis of the jaws: a retrospective study of the background factors and treatment in 104 cases. J Oral Maxillofac Surg. 1997 Jun;55(6):540-4; discussion 545-6. doi: 10.1016/s0278-2391(97)90478-x. PMID 9191633
- [Background] Joseph DL, Shumrick DL. Risks of head and neck surgery in previously irradiated patients. Arch Otolaryngol. 1973 May;97(5):381-4. doi: 10.1001/archotol.1973.00780010393005. No abstract available. PMID 4703530
- [Background] Samuels L, Granick MS, Ramasastry S, Solomon MP, Hurwitz D. Reconstruction of radiation-induced chest wall lesions. Ann Plast Surg. 1993 Nov;31(5):399-405. doi: 10.1097/00000637-199311000-00003. PMID 8285524
- [Background] Hart GB, Mainous EG. The treatment of radiation necrosis with hyperbaric oxygen (OHP). Cancer. 1976 Jun;37(6):2580-5. doi: 10.1002/1097-0142(197606)37:63.0.co;2-h. PMID 949677
- [Background] Marx RE. Osteoradionecrosis: a new concept of its pathophysiology. J Oral Maxillofac Surg. 1983 May;41(5):283-8. doi: 10.1016/0278-2391(83)90294-x. PMID 6572704
- [Background] Marx RE. A new concept in the treatment of osteoradionecrosis. J Oral Maxillofac Surg. 1983 Jun;41(6):351-7. doi: 10.1016/s0278-2391(83)80005-6. No abstract available. PMID 6574217
- [Background] Bevers RF, Bakker DJ, Kurth KH. Hyperbaric oxygen treatment for haemorrhagic radiation cystitis. Lancet. 1995 Sep 23;346(8978):803-5. doi: 10.1016/s0140-6736(95)91620-2. PMID 7674746
- [Background] Woo TC, Joseph D, Oxer H. Hyperbaric oxygen treatment for radiation proctitis. Int J Radiat Oncol Biol Phys. 1997 Jun 1;38(3):619-22. doi: 10.1016/s0360-3016(97)00017-5. PMID 9231688
- [Background] Williams JA Jr, Clarke D, Dennis WA, Dennis EJ 3rd, Smith ST. The treatment of pelvic soft tissue radiation necrosis with hyperbaric oxygen. Am J Obstet Gynecol. 1992 Aug;167(2):412-5; discussion 415-6. doi: 10.1016/s0002-9378(11)91421-5. PMID 1497044
- [Background] Feldmeier JJ, Heimbach RD, Davolt DA, Brakora MJ. Hyperbaric oxygen as an adjunctive treatment for severe laryngeal necrosis: a report of nine consecutive cases. Undersea Hyperb Med. 1993 Dec;20(4):329-35. PMID 8286987